CLINICAL TRIAL: NCT03364062
Title: A Multi-center Study on Effect of Cemented Implantation in Shoulder Replacement on Blood Pressure
Brief Title: Effect of Cemented Implantation in Shoulder Replacement on Blood Pressure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: First Affiliated Hospital of Harbin Medical University (Other); Dalian Medical University (Other); Taoyuan General Hospital (Other Government)
Responsible Party: Principal Investigator, Zhang Peixun, Clinical Professor, Peking University People's Hospital
Other Study IDs: GCS-CISR
Record Dates: First submitted 2017-11-26; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Blood Pressure
Keywords: Blood Pressure; shoulder replacement; proximal humeral fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cemented shoulder replacement patients: A total of 350 cases of proximal humeral fracture receiving cemented shoulder replacement in Department of Orthopedics and Trauma
  Interventions: Procedure: cemented shoulder replacement

INTERVENTIONS:
Procedure: cemented shoulder replacement — proximal humeral fracture receiving hemi-shoulder replacement with cement when inserting the stem

SUMMARY:
To clarify the downward trend of blood pressure affected by bone cement implantation during shoulder replacement operations.

DETAILED DESCRIPTION:
A total of 350 cases of proximal humeral fracture are planned to be recruited and receive semi-shoulder replacement in Department of Orthopedics and Trauma，Peking University People's Hospital．The blood pressure data are collected from patients' anesthesia records. Both the systolic and diastolic blood pressure are recorded at four time spots during operation: the time before using of bone cement (time period A), 0-5 min after using cement (time period B), 5-10 min after using cement (time period C) and 10-15min after using cement (time period D). The data of blood pressure are collected according to anesthesia records．

ELIGIBILITY:
Inclusion Criteria:

•patients with three or four part of proximal humeral fracture receiving cemented shoulder replacement

Exclusion Criteria:

* pathologic fracture
* severe hypertension or hypotension

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with three or four part of proximal humeral fracture, receive shoulder replacement
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-02-10 (Estimated); Primary Completion 2019-12-10 (Estimated); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure | Change from Baseline Systolic Blood Pressure at 15 mins
  the systolic blood pressure after insert the cemented stem

SECONDARY OUTCOMES:
Change from Baseline Diastolic Blood Pressure | Change from Baseline Diastolic Blood Pressure at 15 mins
  the diastolic blood pressure after insert the cemented stem

CONTACTS AND LOCATIONS:
Overall Officials: Yichong Zhang, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No